CLINICAL TRIAL: NCT05687552
Title: Role of 18F-FDG PET/CT in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Saber Ahmed, assisstant lecturer, Sohag University
Other Study IDs: gastric cancer
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pet -ct — assessment of added value of pet -ct in patients with gastric cancer and how patient get benefit from this finding

SUMMARY:
The objective of the study is to assess the value of PET/CT in diagnosis, staging, response evaluation, and relapse monitoring of gastric cancer.

DETAILED DESCRIPTION:
gastric cancer (GC) is the fifth most common malignancy and the third leading cause of cancer mortality worldwide (1) It carries a poor prognosis, with a 5-year survival of only 20%-30% (2) Clinical staging, based mainly on imaging, is critical in determining the best treatment.There is a widely accepted consensus of the usefulness of FDG PET/CT in staging and restaging of gastric cancer. According to evidence-based data, this modality can evaluate gastric cancer more accurately and is helpful for evaluation of tumor biologic characteristics, detection of lymph node and distant metastases, assessment of tumor response to therapy(9).

retrospective and prospective study will conducted at Sohag oncology hospital, nuclear medicine unit& Assuit university hospital, nuclear medicine unit including 50 patients in 12 months .

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed as GC on surgically resected specimens;
2. Patients with gastric and extragastric metastasis.
3. patients with gastric cancer either operated or not.

Exclusion Criteria:

1. Patients with second malignancy.
2. Patient without proven pathology of cancer stomach.
3. Severely ill patient (patient with disturbed conscious level, or couldn't lay supine during the imaging).
4. uncontrolled diabetic patient with blood glucose level more than 200mg\dl.
5. pregnant women

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient diagnosed by pathology as gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
comparison of pet -ct finding with ct finding | base line
  The 18F-FDG PET/CT scan is visually estimated in the patients included in the study and quantitatively assessed by estimation of standardized uptake value(suv max). Statistical analysis of the included quantitative data.

CONTACTS AND LOCATIONS:
Overall Officials: wafaa elmaghraby, ass prof, Study Director — Sohag University; mohamed soliman, prof, Study Director — Sohag University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang L, Wang XJ, Baba H, Giganti F. Gastric cancer and image-derived quantitative parameters: Part 2-a critical review of DCE-MRI and 18F-FDG PET/CT findings. Eur Radiol. 2020 Jan;30(1):247-260. doi: 10.1007/s00330-019-06370-x. Epub 2019 Aug 7. PMID 31392480
- [Background] Saka M, Katai H, Fukagawa T, Nijjar R, Sano T. Recurrence in early gastric cancer with lymph node metastasis. Gastric Cancer. 2008;11(4):214-8. doi: 10.1007/s10120-008-0485-4. Epub 2009 Jan 8. PMID 19132483
- [Result] Liu Q, Li J, Xin B, Sun Y, Feng D, Fulham MJ, Wang X, Song S. 18F-FDG PET/CT Radiomics for Preoperative Prediction of Lymph Node Metastases and Nodal Staging in Gastric Cancer. Front Oncol. 2021 Sep 13;11:723345. doi: 10.3389/fonc.2021.723345. eCollection 2021. PMID 34589429